CLINICAL TRIAL: NCT03870516
Title: Assessment of Subclinical Left Atrial and Left Ventricular Dysfunction by Speckle Tracking Echocardiography in Severe Asymptomatic Rheumatic Mitral Regurgitation and Its Role in Predicting Outcome After Valve Replacement Compared to Guideline Parameters
Brief Title: Left Chamber Function in Mitral Regurgitation and Predicting Outcome After Replacement and Targeting for Early Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed M. Reda Abdelaziz, physician, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Speckle tracking echo
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Mitral Regurgitation
Keywords: mitral; regurgitation; speckle; echocardiography; replacement
MeSH Terms: conditions — Mitral Valve Insufficiency; Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Patients with rheumatic severe mitral regurgitation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Valve replacement according to guideline parameters (Placebo Comparator): One group will be referred for surgery according according to indications for mitral valve replacement in European guidelines for valvular heart diseases published in 2017 and will have speckle tracking echocardiography before surgery and 6 months later for comparison.
  Interventions: Procedure: Mitral valve replacement; Device: Speckle tracking echocardiography
- Early valve replacement (Active Comparator): The other group will include patients with severe asymptomatic mitral regurgitation who have left atrial or left ventricular dysfunction according to speckle tracking echocardiography and will be referred to surgery, then speckle tracking echo will be performed 6 months later.
  Interventions: Procedure: Mitral valve replacement; Device: Speckle tracking echocardiography

INTERVENTIONS:
Procedure: Mitral valve replacement — Replacing the diseased mitral valve in cases with severe mitral regurgitation with a prosthetic valve.
Device: Speckle tracking echocardiography — We will perform Speckle tracking echocardiography in order to identify patients with early subclinical left ventricular or left atrial dysfunction and refer them to surgery, Then after surgery, speckle tracking echocardiography will be performed for all patients to assess improvement of left atrial (conduit, reservoir and booster contractile functions) and left ventricular (global longitudinal strain) function

SUMMARY:
The study aims to analyze the role of left ventricular and left atrial functional parameters by speckle tracking echocardiography in predicting outcome after mitral valve replacement and targeting for early intervention compared to guideline parameters.

DETAILED DESCRIPTION:
Without surgical treatment, the 10-year morbidity and mortality for patients with severe mitral regurgitation can be as high as 90%.

In contrast, with successful surgical correction of mitral regurgitation before the appearance of symptoms, patients may have life expectancies similar to that of the general population.

According to European recommendations, mitral valve replacement must be proposed to symptomatic patients and to patients with significant left ventricular remodeling as a consequence of the severity of mitral regurgitation.

A significant decline in left ventricular function is defined, in these recommendations, echocardiographically as an left ventricular ejection fraction < 60% or an left ventricular end-systolic diameter > 45 mm.

Preoperative left ventricular systolic function and left ventricular end systolic diameter are important postoperative prognostic factors.

The early detection of left ventricular systolic dysfunction remains a challenge. Mitral regurgitation causes low left ventricular afterload, and the ejection fraction thus remains normal or supernormal until the disease reaches an advanced stage.

Some authors have suggested the additive value of deformation indices as more sensitive than the ejection fraction to detect subclinical left ventricular systolic dysfunction Speckle tracking echocardiography has been well validated as a quantitative assessment tool for left ventricular function, and more recently this technique has been described for assessment of regional and global left atrial function

ELIGIBILITY:
Inclusion Criteria:

* Patients with rheumatic severe mitral regurgitation who will have mitral valve replacement in Assiut University Heart Hospital

Exclusion Criteria:

* Degenerative mitral regurgitation, ischemic mitral regurgitation, severe rheumatic mitral regurgitation with atrial fibrillation or impaired left ventricular ejection fraction, associated mitral stenosis, or significant aortic regurgitation and ischemic heart disease.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-20 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Recovery of left atrial functions (conduit, reservoir and booster contractile functions) and left ventricular function (global longitudinal strain) by speckle tracking echocardiography after mitral valve replacement | 6 months after surgery
  Speckle tracking echocardiography will be performed 6 months after surgery to assess recovery of left atrial function by assessment of conduit, reservoir and booster contractile functions and left ventricular function by assessment of global longitudinal strain after mitral valve replacement

SECONDARY OUTCOMES:
Number of patients with major adverse cardiovascular events (MACE) | 6 months
  Quantifying patients with CVD events, admission for HF, ischemic cardiovascular events, cardiac death, or MACE within 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy Shamseddin, PhD, Study Chair — Assiut University

REFERENCES:
- [Background] Lancellotti P, Cosyns B, Zacharakis D, Attena E, Van Camp G, Gach O, Radermecker M, Pierard LA. Importance of left ventricular longitudinal function and functional reserve in patients with degenerative mitral regurgitation: assessment by two-dimensional speckle tracking. J Am Soc Echocardiogr. 2008 Dec;21(12):1331-6. doi: 10.1016/j.echo.2008.09.023. PMID 19041577
- [Background] Marciniak A, Sutherland GR, Marciniak M, Kourliouros A, Bijnens B, Jahangiri M. Prediction of postoperative left ventricular systolic function in patients with chronic mitral regurgitation undergoing valve surgery--the role of deformation imaging. Eur J Cardiothorac Surg. 2011 Nov;40(5):1131-7. doi: 10.1016/j.ejcts.2011.02.049. Epub 2011 Apr 1. PMID 21459016
- [Background] Vianna-Pinton R, Moreno CA, Baxter CM, Lee KS, Tsang TS, Appleton CP. Two-dimensional speckle-tracking echocardiography of the left atrium: feasibility and regional contraction and relaxation differences in normal subjects. J Am Soc Echocardiogr. 2009 Mar;22(3):299-305. doi: 10.1016/j.echo.2008.12.017. PMID 19258177
- [Background] Cameli M, Caputo M, Mondillo S, Ballo P, Palmerini E, Lisi M, Marino E, Galderisi M. Feasibility and reference values of left atrial longitudinal strain imaging by two-dimensional speckle tracking. Cardiovasc Ultrasound. 2009 Feb 8;7:6. doi: 10.1186/1476-7120-7-6. PMID 19200402